CLINICAL TRIAL: NCT01614249
Title: Role of Omega-3 Fish Oil Fatty Acids on Depression Among HIV-seropositive Pregnant Pregnant Women in Nairobi: A Randomized Double-blind Controlled Trial
Brief Title: Omega-3 Supplementation and Depression Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: Consortium for Advanced Research Training in Africa (CARTA) (Unknown); Innovix Pharma Inc. (Unknown)
Responsible Party: Principal Investigator, Rose Okoyo Opiyo, Principal Investigator (PI), University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ODR-2011/2012; ECCT/12/03/01 (Registry Identifier: Pharmacy and Poisons Board, Kenya)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Depressive Symptoms
Keywords: Omega-3; EPA; Depression; HIV infected; Pregnant women
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soybean oil soft gels (Placebo Comparator): Participants on this arm will receive a dietary supplement of OmegaVia soybean oil soft gels as a placebo for 8 weeks with bi-weekly follow-up visits to monitor side effects and compliance.
  Interventions: Dietary Supplement: Soybean oil soft gels
- Fish oil omega-3 EPA-rich soft gels (Experimental): Participants will receive OmegaVia fish oil omega-3 EPA-rich soft gels to take orally for eight (8) weeks with bi-weekly follow-up visits for monitoring of side effects and compliance and data collection.
  Interventions: Dietary Supplement: Fish oil omega-3 EPA-rich soft gels

INTERVENTIONS:
Dietary Supplement: Soybean oil soft gels — Each participant will receive OmegaVia soybean oil soft gels to take orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks
  Other Names: OmegaVia Soybean oil soft gels
  Arms: Soybean oil soft gels
Dietary Supplement: Fish oil omega-3 EPA-rich soft gels — A total of 3.0g of OmegaVia fish oil omega-3 EPA-rich soft gels will be taken orally per day as one soft gel in the morning, mid-day and evening after meals for 8 weeks with bi-weekly follow-up visits.
  Other Names: OmegaVia fish oil omega-3 EPA-rich soft gels
  Arms: Fish oil omega-3 EPA-rich soft gels

SUMMARY:
Fish oil omega-3 supplements provide essential nutrients for brain health and functioning. These nutrients have been proven to be effective in reducing depressive symptoms. They have also been found to be effective and well tolerated in reducing the bad fat accumulation among patients infected with human immunodeficiency virus (HIV)and are using highly active antiretroviral treatment. The role of this nutritional supplement in combating depression among pregnant women who are living with HIV infection has however not been established. Yet, currently, more than 2 million pregnant women are estimated to be living with HIV infection globally. In Kenya, about 9.0% of pregnant women are HIV-seropositive.

In this study, it is hypothesized that there is no difference in the levels of depressive symptoms among HIV infected pregnant women who are taking omega-3 fish oil supplements and those taking a placebo.

The study will therefore seek to ascertain that taking omega-3 fish oil nutritional supplement has a significant positive effect on depressive symptoms among HIV infected pregnant women, compared to a placebo.

DETAILED DESCRIPTION:
Background to the study: Fatty acids are the key building blocks of most fats and oils, both those in the body and in foods. Among the essential fatty acids that are required to maintain health, but must come from the diet, is omega-3. These omega-3 fatty acids are important constituents of all cell membranes and are involved in the movement of substances in and out of the cells. They also produce hormone-like substances which regulate many functions of the body. The omega-3 fatty acids occur naturally, and consist of shorter long-chain alphalinolenic acid (ALA) and the longer chain, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). The ALA is naturally found in green leafy vegetables, flax seed, soybean oil and walnuts. The long chain EPA and DHA are naturally found in dark muscles of sea fish such as salmon, mackerel and tuna. These nutrients must be consumed in the diet because they cannot be synthesized by humans[1]. Research on the health benefits of omega-3 fatty acids dates back to 1929 when it was found to promote growth and prevent inflammation of the skin in rats [2, 3]. The essentiality of long-chain fatty acids for human health however emerged in 1970's when the first total parenteral nutrition which was fat-free was found to induce the essential fatty acid deficiencies among infants with volvulus, a bowel obstruction, at birth[4]. Further research in the 1970s on the health status of modern-hunter-gatherer Inuit Eskimos was also found to be related to their staple diet of fatty sea fish and fish eating marine mammals rich in long chain omega-3 fatty acids, EPA and DHA [5].

It has been proven that omega-3 long chain fatty acids, EPA and DHA improve depressive symptoms [6, 7]. As a mood disorder, depression is characterized by feelings of unhappiness and hopelessness, and generally marked by altered mood. It is not a single disease, but a syndrome encompassing a spectrum of symptoms with multiple causes [8, 9]. Women experience at least one episode of minor or major depression during pregnancy and after childbirth. This is however often under-diagnosed, undetected and missed out due to lack of screening. Although screening for depression may not be a routine activity in antenatal care, studies that have screened for depression in pregnancy indicate that 20-30% of pregnant women are depressed [10, 11]. The prevalence of depression is high during the second and third trimesters of pregnancy [12] when maternal level of omega-3 fatty acids is depleted.

Adequate intake of long chain omega-3 fatty acids is also essential, during pregnancy to support normal growth and maturation of many fetal organ systems, particularly the brain and eyes [13, 14]. Moreover, long chain omega-3 fatty acids are critical for the development and function of many different organ systems of the fetus, including the structure of the brain and retina of the eye [15]. Premature birth and its potential neurological complications may result from omega-3 deficiency [16]. Documented research findings on omega-3 fatty acids and human immune-deficiency virus/ acquired immunodeficiency syndrome (HIV/AIDS) are mainly two-fold: one, on plasma triglycerides levels, and two, on the immune response parameters. Studies have shown that use of omega-3 fatty acids among HIV infected patients receiving highly active antiretroviral therapy is well tolerated and effective in reducing the plasma triglyceride levels [17-19]. The fish oil has therefore been recommended as second-line therapy for HIV patients with hypertriglyceridemia [12]. One of the metabolic end products of long chain fatty acids of omega-3 and omega-6, once eaten and absorbed by the body, are prostaglandin hormones which are responsible for the inflammation response. Research shows that omega-3 fatty acids produce less prostaglandin than omega-6 fatty acids, decreasing the inflammatory process [5]. Earlier research reported that omega-3 fish oil is immuno-suppressive as it significantly decreased various parameters of the immune response [20]. However, more recent studies have shown that dietary intake of omega-3 fatty acids increased the cluster of differentiation 4 (CD4) cell count [21] The role of long chain omega-3 fatty acids in combating depression among HIV-seropositive pregnant women has however not been established. The specific symptoms which may be more responsive to omega-3 supplementation have also not been established. Currently, more than 2 million pregnant women are estimated to be living with HIV infection globally. In Kenya, about 9.0% of pregnant women are HIV-seropositive [22] and their health conditions as well as that of their unborn babies silently continue to deteriorate partly due to depression related comorbidities. This research will seek to ascertain that taking omega-3 fish oil supplement with higher EPA in relation to DHA can have a significant positive effect on depressive symptoms among HIV-seropositive pregnant women compared to a placebo. It will also monitor and identify those depressive symptoms that are more responsive to this nutrient among the HIV-seropositive pregnant women, and can be managed through nutrition supplementation.

Conceptual Framework: The major risk factors for depression are genetic predisposition, hormonal imbalance and stressful events which could be of environmental, social or psychological origin as well as nutrition-related factors [11, 23-25]. Stressful events could however also cause hormonal imbalance, which, in the process can increase the stress hormone, cortisol, causing depression [23]. Both pregnancy and HIV infection status are also accompanied by high nutrient demand, in the presence of inadequate and inappropriate dietary intake as well as a high intake of saturated fats in fried food. This is likely to contribute to nutrient deficiencies, which also determines the neurotransmitter function and hormonal balance in mental health.

Problem statement: This study seeks to ascertain that taking omega-3 fish oil supplement with higher EPA in relation to DHA have a significant positive effect on depressive symptoms among HIV-seropositive pregnant women. The level of omega-3 fatty acids rapidly declines during pregnancy as some of it is transferred to the fetus for the rapid formation of the fetal brain cells [13]. The resultant depletion in omega-3 might precipitate the occurrence of depression in pregnant women unless the nutrient deficit is met through dietary intake of omega-3 rich foods or supplementation. The modern diet is however inadequate in long chain omega-3 fatty acids [5]. About 40% of HIV-seropositive pregnant women are reportedly depressed [26, 27]. The depression in HIV-seropositive pregnant women is a significant public health problem due to its negative effects on both maternal and child health. It may adversely affect the quality of life and adherence to HIV/AIDS medication regimens [27, 28] which may subsequently affect disease progression and health outcome [29] of the women. Currently, more than 2 million pregnant women are estimated to be living with HIV infection globally [9]. In Kenya, about 9.0% of pregnant women are HIV-seropositive [22].

Justification of the study: This study will contribute to the debate on nutritional support and management of depressive symptoms and related health complications in HIV infected pregnant women and other vulnerable populations, to improve their mental health, hence improve the quality of life. A reduction in the prevalence of depression could therefore influence nutrition and health agencies as well as policy makers to make omega-3 fatty acid nutritional supplement accessible to HIV positive pregnant women and other vulnerable populations.

Overall aim: To ascertain that taking omega-3 fish oil supplement with higher EPA in relation to DHA have a significant positive effect on depressive symptoms compared to a placebo among HIV-seropositive pregnant women.

Research questions: 1.Does taking omega-3 fish oil supplement with higher EPA in relation to DHA have a significant positive effect on depressive symptoms among HIV-seropositive pregnant women, compared to a placebo? 2. Is the change in depressive symptom levels among study participants related to the change in their omega-3 fatty acid status after intervention with omega-3 fish oil supplement and placebo? 3. Which depressive symptoms are more responsive to omega-3 fish oil supplement intervention?

Study setting: The study will be conducted at health facilities in Nairobi, Kenya. According to the latest Kenya national population and housing census results of 2009, [30], Nairobi, which is the capital city of Kenya, is the most populated city in the country with about 3.1 million people (about 1.6 million males and 1.5 million females) and an annual growth rate of about 4.1%[16]. The available sentinel survey data indicate that the prevalence of HIV/AIDS among pregnant women in Nairobi was 10.1% [31] in 2006.

Methodology: This will be a double-blind, parallel randomized control trial (RCT) using omega-3 fish oil supplements and placebo. Both the study participants and the research administrators, including the principle investigator, will not know the difference between omega-3 supplement and placebo which will be of similar physical characteristics. Participants will be recruited from purposely sampled health facilities with highest attendance at the Prevention-of Mother-to-Child-Transmission (PMTCT) of HIV AIDS programs. The sampling frame will consist of pregnant women with known HIV-seropositive status and enrolled in PMTCT program at these health facilities. A total of 200 women who meet the study inclusion and exclusion criteria will be enrolled to participate in the study.

Data Collection: Quantitative methods will be used to collect socio-demographic information, dietary intake data, and depressive symptoms, biological specimens of cheek cells, maternal weight, CD4 count, blood pressure and compliance with routine medication and study intervention. The primary measurement tool for efficacy of omega-3 fish oil will be the Beck Depression Inventory, Second Edition (BDI-II) scoring scale with a cut-off score for depression of 14 or more. Further understanding of depression in pregnancy and HIV/AIDS condition will be gained through qualitative methods. Cheek cell samples will be collected through mouth wash method for laboratory extraction of lipids for omega-3 analysis. The lipids will be extracted from the cheek cells using Bligh and Dyer methodology [32]. Gas-liquid chromatography by the method of Gibson and Kneebone [33] will be used to determine per cent (%) levels of omega-3 fatty acids in the lipids before, during and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant HIV seropositive women with known CD4 cell count less than 500
* Pregnant women who are in their 2nd trimester of pregnancy (Week 13-27).
* Normal nutritional status pregnancy with mid-upper arm circumference (MUAC of 22 cm - 33 cm)at entry into the study;
* Beck Depression Inventory Second Edition (BDI-II) Scale scores at entry into the study of 14 or more;
* Pregnant HIV positive women who will give consent to participate in the study

Exclusion Criteria:

* Underweight with MUAC less than 22 cm and overweight with MUAC more than 33 cm at entry into the study;
* Pregnant women taking antidepressant medications;
* Those on anti-clotting medication (those with liver disease, varicose veins, peptic ulcers); or Vitamin K supplement. Omega-3 supplements may increase their effects;
* Those on diabetic medication since Omega-3 may increase their blood sugar.
* Incomplete depression screening form (more than 5 items unanswered)
* Those whose BDI-II screening scores are less than 14;
* Those women currently taking omega-3 nutritional supplement
* Pregnant HIV-seropositive women without consent to participate in the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose O. Opiyo, MSc, Principal Investigator — University of Nairobi
Locations (1):
- Nairobi City Council Health Facilities, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data available on request

REFERENCES:
- [Background] Jones, P. and A. Papamandjaris, eds. Lipid: Cellular Metabolism in Present Knowledge in Nutrition. 8th ed. Present Knowledge in Nutrition, ed. B. Bowman and R. Russell2001, ILSI Press: Washington, DC. 104-114.
- [Background] Burr GO, Burr MM. Nutrition classics from The Journal of Biological Chemistry 82:345-67, 1929. A new deficiency disease produced by the rigid exclusion of fat from the diet. Nutr Rev. 1973 Aug;31(8):248-9. doi: 10.1111/j.1753-4887.1973.tb06008.x. No abstract available. PMID 4586201
- [Background] Holman RT. The slow discovery of the importance of omega 3 essential fatty acids in human health. J Nutr. 1998 Feb;128(2 Suppl):427S-433S. doi: 10.1093/jn/128.2.427S. PMID 9478042
- [Background] Paulsrud JR, Pensler L, Whitten CF, Stewart S, Holman RT. Essential fatty acid deficiency in infants induced by fat-free intravenous feeding. Am J Clin Nutr. 1972 Sep;25(9):897-904. doi: 10.1093/ajcn/25.9.897. No abstract available. PMID 4626563
- [Background] Stoll, A., The Omega-3 connection.2001, New York.: Simon & Schuster.
- [Background] Lesperance F, Frasure-Smith N, St-Andre E, Turecki G, Lesperance P, Wisniewski SR. The efficacy of omega-3 supplementation for major depression: a randomized controlled trial. J Clin Psychiatry. 2011 Aug;72(8):1054-62. doi: 10.4088/JCP.10m05966blu. Epub 2010 Jun 15. PMID 20584525
- [Background] Panagiotakos DB, Mamplekou E, Pitsavos C, Kalogeropoulos N, Kastorini CM, Papageorgiou C, Papadimitriou GN, Stefanadis C. Fatty acids intake and depressive symptomatology in a Greek sample: an epidemiological analysis. J Am Coll Nutr. 2010 Dec;29(6):586-94. doi: 10.1080/07315724.2010.10719897. PMID 21677122
- [Background] Leung BM, Kaplan BJ. Perinatal depression: prevalence, risks, and the nutrition link--a review of the literature. J Am Diet Assoc. 2009 Sep;109(9):1566-75. doi: 10.1016/j.jada.2009.06.368. PMID 19699836
- [Background] WHO/UNAIDS/UNICEF, Towards Universal Access: Scaling up priority HIV/AIDS interventions in the health sector. Progress Report, April 2007., 2007.
- [Background] Goodman JH, Tyer-Viola L. Detection, treatment, and referral of perinatal depression and anxiety by obstetrical providers. J Womens Health (Larchmt). 2010 Mar;19(3):477-90. doi: 10.1089/jwh.2008.1352. PMID 20156110
- [Background] Marcus SM, Flynn HA, Blow FC, Barry KL. Depressive symptoms among pregnant women screened in obstetrics settings. J Womens Health (Larchmt). 2003 May;12(4):373-80. doi: 10.1089/154099903765448880. PMID 12804344
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Hornstra G. Essential fatty acids in mothers and their neonates. Am J Clin Nutr. 2000 May;71(5 Suppl):1262S-9S. doi: 10.1093/ajcn/71.5.1262s. PMID 10799400
- [Background] Innis SM, Friesen RW. Essential n-3 fatty acids in pregnant women and early visual acuity maturation in term infants. Am J Clin Nutr. 2008 Mar;87(3):548-57. doi: 10.1093/ajcn/87.3.548. PMID 18326591
- [Background] Melina, V. and B. Davis, The New Becoming Vegetarian. The essential guide to a healthy vegetarian diet. 2003, Tennessee: Healthy Living Publications.
- [Background] Cetin I, Koletzko B. Long-chain omega-3 fatty acid supply in pregnancy and lactation. Curr Opin Clin Nutr Metab Care. 2008 May;11(3):297-302. doi: 10.1097/MCO.0b013e3282f795e6. PMID 18403927
- [Background] Carter VM, Woolley I, Jolley D, Nyulasi I, Mijch A, Dart A. A randomised controlled trial of omega-3 fatty acid supplementation for the treatment of hypertriglyceridemia in HIV-infected males on highly active antiretroviral therapy. Sex Health. 2006 Dec;3(4):287-90. doi: 10.1071/sh06001. PMID 17112442
- [Background] Gerber JG, Kitch DW, Fichtenbaum CJ, Zackin RA, Charles S, Hogg E, Acosta EP, Connick E, Wohl D, Kojic EM, Benson CA, Aberg JA. Fish oil and fenofibrate for the treatment of hypertriglyceridemia in HIV-infected subjects on antiretroviral therapy: results of ACTG A5186. J Acquir Immune Defic Syndr. 2008 Apr 1;47(4):459-66. doi: 10.1097/QAI.0b013e31815bace2. PMID 17971707
- [Background] Wohl DA, Tien HC, Busby M, Cunningham C, Macintosh B, Napravnik S, Danan E, Donovan K, Hossenipour M, Simpson RJ Jr. Randomized study of the safety and efficacy of fish oil (omega-3 fatty acid) supplementation with dietary and exercise counseling for the treatment of antiretroviral therapy-associated hypertriglyceridemia. Clin Infect Dis. 2005 Nov 15;41(10):1498-504. doi: 10.1086/497273. Epub 2005 Oct 11. PMID 16231263
- [Background] Meydani SN, Lichtenstein AH, Cornwall S, Meydani M, Goldin BR, Rasmussen H, Dinarello CA, Schaefer EJ. Immunologic effects of national cholesterol education panel step-2 diets with and without fish-derived N-3 fatty acid enrichment. J Clin Invest. 1993 Jul;92(1):105-13. doi: 10.1172/JCI116537. PMID 8325975
- [Background] de Luis DA, Bachiller P, Izaola O, Eiros Bouza JM. [Relation between intake of omega 3 fatty acids and CD4 count in patients with HIV infection: a transversal study]. An Med Interna. 2005 Jul;22(7):323-5. Spanish. PMID 16288576
- [Background] NASCOP, Kenya AIDS Indicator Survey, (KAIS) 2007, 2009, NASCOP: Nairobi. p. 11.
- [Background] Kammerer M, Taylor A, Glover V. The HPA axis and perinatal depression: a hypothesis. Arch Womens Ment Health. 2006 Jul;9(4):187-96. doi: 10.1007/s00737-006-0131-2. Epub 2006 May 19. PMID 16708167
- [Background] Thase ME. The role of neurobiologic processes in symptoms of depression. J Clin Psychiatry. 2011 Feb;72(2):e08. doi: 10.4088/JCP.9078tx3c. PMID 21382303
- [Background] Warner R, Appleby L, Whitton A, Faragher B. Demographic and obstetric risk factors for postnatal psychiatric morbidity. Br J Psychiatry. 1996 May;168(5):607-11. doi: 10.1192/bjp.168.5.607. PMID 8733800
- [Background] Ickovics JR, Hamburger ME, Vlahov D, Schoenbaum EE, Schuman P, Boland RJ, Moore J; HIV Epidemiology Research Study Group. Mortality, CD4 cell count decline, and depressive symptoms among HIV-seropositive women: longitudinal analysis from the HIV Epidemiology Research Study. JAMA. 2001 Mar 21;285(11):1466-74. doi: 10.1001/jama.285.11.1466. PMID 11255423
- [Background] Smith Fawzi MC, Kaaya SF, Mbwambo J, Msamanga GI, Antelman G, Wei R, Hunter DJ, Fawzi WW. Multivitamin supplementation in HIV-positive pregnant women: impact on depression and quality of life in a resource-poor setting. HIV Med. 2007 May;8(4):203-12. doi: 10.1111/j.1468-1293.2007.00454.x. PMID 17461847
- [Background] Cook JA, Cohen MH, Burke J, Grey D, Anastos K, Kirstein L, Palacio H, Richardson J, Wilson T, Young M. Effects of depressive symptoms and mental health quality of life on use of highly active antiretroviral therapy among HIV-seropositive women. J Acquir Immune Defic Syndr. 2002 Aug 1;30(4):401-9. doi: 10.1097/00042560-200208010-00005. PMID 12138346
- [Background] Cruess DG, Douglas SD, Petitto JM, Have TT, Gettes D, Dube B, Cary M, Evans DL. Association of resolution of major depression with increased natural killer cell activity among HIV-seropositive women. Am J Psychiatry. 2005 Nov;162(11):2125-30. doi: 10.1176/appi.ajp.162.11.2125. PMID 16263853
- [Background] KNBS, Kenya 2009 Population and Housing Census, M.o.P.a.N. Development, Editor 2010, Government Printers: Nairobi.
- [Background] NASCOP/MOH/CDC, Sentinel Surveillance of HIV & STDs in Kenya Report 2006, 2006, NASCOP: Nairobi.
- [Background] BLIGH EG, DYER WJ. A rapid method of total lipid extraction and purification. Can J Biochem Physiol. 1959 Aug;37(8):911-7. doi: 10.1139/o59-099. No abstract available. PMID 13671378
- [Background] Gibson RA, Kneebone GM. Effect of sampling on fatty acid composition of human colostrum. J Nutr. 1980 Aug;110(8):1671-5. doi: 10.1093/jn/110.8.1671. PMID 7400857
- [Derived] Opiyo RO, Nyasulu PS, Koigi RK, Obondo A, Ogoyi D, Kogi-Makau W. Effect of fish oil omega-3 fatty acids on reduction of depressive symptoms among HIV-seropositive pregnant women: a randomized, double-blind controlled trial. Ann Gen Psychiatry. 2018 Nov 26;17:49. doi: 10.1186/s12991-018-0220-4. eCollection 2018. PMID 30534187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women who met the trial inclusion criteria were recruited from clinic registers at their respective Prevention of mother-to-child transmission program clinics from July 2012 to May 2013 with assistance from mentor-mothers in the clinics. Women visiting the clinics first time were included in clinic registers and invited to participate in the trial.
Pre-assignment Details: Participants were assigned to either of the trial arms soon after enrollment to minimize drop-outs which might have occurred if enrolled participants exceeded gestation age or gave birth before randomization.
Groups:
- Soybean Oil Soft Gels Control Group: As a control group, participants received OmegaVia soybean oil soft gels for eight weeks with regular cell-phone and bi-weekly face-to-face follow-up visits. During each follow-up visit, participants were re-supplied with soft-gels and monitored for side effects and compliance.
  Each participant randomly received a sequentially numbered, securely sealed opaque plastic bottle containing soybean oil soft gels to take for two weeks before returning for re-supply. Three soft gels of soybean oil were taken by each participant per day. Each soft gel contained saturated fatty acids (0.178 grams), monounsaturated fatty acids (0.299 grams) and polyunsaturated fatty acids (0.985 grams) with traces of eicosapentaenoic acid (EPA), of 0.115 grams. The soft gels were taken orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks.
- Fish Oil Omega-3 EPA-rich Experimental Group: As the experimental group, participants received dietary supplement of OmegaVia fish oil omega-3 EPA-rich soft gels to take orally for eight weeks with bi-weekly follow-up visits. During each follow-up visit, participants were re-supplied with soft-gels and monitored for side effects and compliance.
  Each participant randomly received a sequentially numbered, securely sealed opaque plastic bottle containing fish oil omega-3 EPA-rich soft gels to take for two weeks before returning for re-supply. Three soft gels of fish oil omega-3 fatty acid were taken by each participant per day. Each soft gel contained more eicosapentaenoic acid (EPA) of 0.715 grams than docosahexaenoic acid (DHA) of 0.340 grams. The soft gels were taken orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks.
Period: Overall Study
Arm/Group | Soybean Oil Soft Gels Control Group | Fish Oil Omega-3 EPA-rich Experimental Group
Started | 107 (Participants received every two-weeks supply and monitored regularly on cell-phone and face-to-face.) | 109 (Participants received every two-week supply and monitored regularly on cell-phone and face-to-face.)
At Week-4 | 98 (Participants received every two-week supply and monitored regularly on cell-phone and face-to-face.) | 92 (Participants received every two-week supply and monitored regularly on cell-phone and face-to-face.)
At Week-8 (End of Study Period) | 96 (End of study data collected for all participants who completed the 8-week trial period.) | 86 (End of study data collected for all participants who completed the 8-week trial period.)
Completed | 96 (End of study data analyzed for only participants who completed the 8-week trial period.) | 86 (End of study data analyzed for only participants who completed the 8-week trial period.)
Not Completed | 11 | 23
Not completed — Lost to Follow-up | 11 | 23

BASELINE CHARACTERISTICS:
Groups:
- Fish Oil Omega-3 EPA-rich Soft Gels Experimental Group: As the intervention group, participants received a dietary supplement of Omega Via fish oil omega-3 EPA-rich soft gels to take orally for eight weeks with bi-weekly follow-up visits to resupply the soft-gels, monitoring of side effects and compliance and data collection.
  Each participant randomly received a sequentially numbered, securely sealed opaque plastic bottle containing fish oil omega-3 EPA-rich soft gels to take for two weeks before returning for re-supply. Each participants took three soft gels of fish oil omega-3 fatty acid per day, each containing more EPA (0.715 grams) than docosahexaenoic acid (DHA) of 0.340 grams. The soft gels were taken orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Soybean Oil Soft Gels Control Group | Fish Oil Omega-3 EPA-rich Soft Gels Experimental Group | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 10
  Between 18 and 65 years | 102 | 104 | 206
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 26 [22 to 30] | 26 [22 to 30] | 26 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 216
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 107 | 109 | 216
Gestation age [Median (Inter-Quartile Range); unit: Weeks] | 22 [19 to 24] | 22 [18 to 24] | 22 [18 to 24]
Cluster of differentiation 4 (CD4) cell count [Median (Inter-Quartile Range); unit: cells/µl] | 360 [288 to 414] | 361 [287 to 440] | 360 [288 to 425]
Mid-upper-arm circumference (MUAC) [Median (Inter-Quartile Range); unit: cm] | 26.0 [24.3 to 28.0] | 26.0 [23.9 to 27.6] | 26.0 [24.0 to 27.8]
BDI-II depressive symptom scores [Median (Inter-Quartile Range); unit: Scores on a scale] — Beck Depression Inventory Second Edition (BDI-II) Scale is a 21-item scoring tool which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represent a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe).Scores for each symptom are added up to obtain the total scores for all 21 items, which are interpreted as follows: Scores of 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression and 29-63: severe depression.
  Scores on a scale | 21 [17 to 25] | 20 [16 to 25] | 21 [17 to 25]
Marital status [Number; unit: participants]
  Single (not married, divorced, widowed | 22 | 27 | 49
  Married | 85 | 82 | 167
Parity [Number; unit: participants]
  First pregnancy | 24 | 24 | 48
  Not first pregnancy | 83 | 85 | 168
Education status [Number; unit: participants]
  No High school education | 55 | 55 | 110
  At least High school education | 52 | 54 | 106
Employment status [Number; unit: participants]
  Not in gainful employment | 64 | 61 | 125
  In gainful employment with income | 43 | 48 | 91
Household income per month [Median (Inter-Quartile Range); unit: Kenya Shillings (Ksh.)] | 5025 [3000 to 8000] | 6000 [3000 to 8000] | 5050 [3000 to 8000]
HIV status knowledge before pregnancy [Number; unit: participants]
  No, newly tested less than 6 months | 56 | 56 | 112
  Yes, known positive, 6 months plus | 51 | 53 | 104
HIV status disclosure to anyone [Number; unit: participants]
  Not disclosed | 25 | 18 | 43
  Disclosed to someone | 82 | 91 | 173
prevention of mother-to-child transmission program m2m support group meeting attendance [Number; unit: participants]
  Not attended | 54 | 62 | 116
  Attended | 53 | 47 | 100
Experienced stressful life event [Number; unit: participants]
  None 2 weeks before study | 75 | 73 | 148
  Yes, 2 weeks before study | 32 | 36 | 68
Dietary vitamin C [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 59 | 62 | 121
  At least EAR for pregnant women | 48 | 47 | 95
Dietary vitamin B1 [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 67 | 73 | 140
  At least EAR for pregnant women | 40 | 36 | 76
Dietary vitamin B6 [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 87 | 85 | 172
  At least EAR for pregnant women | 20 | 24 | 44
Dietary vitamin B12 [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 94 | 97 | 191
  At least EAR for pregnant women | 13 | 12 | 25
Dietary folate [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 91 | 98 | 189
  At least EAR for pregnant women | 16 | 11 | 27
Dietary Iron [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 107 | 109 | 216
  At least EAR for pregnant women | 0 | 0 | 0
Dietary vitamin E [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 87 | 89 | 176
  At least EAR for pregnant women | 20 | 20 | 40
Dietary calcium [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 79 | 78 | 157
  At least EAR for pregnant women | 28 | 31 | 59
Dietary selenium [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 76 | 82 | 158
  At least EAR for pregnant women | 31 | 27 | 58
Dietary zinc [Number; unit: participants]
  Below Estimated Average Requirement (EAR) | 105 | 109 | 214
  At least EAR for pregnant women | 2 | 0 | 2
Dietary total omega-3 [Number; unit: participants]
  Below Recommended daily intake | 89 | 99 | 188
  At least recommended daily intake | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in BDI-II Depressive Symptom Scores
Description: Depressive symptoms were assessed by Beck Depression Inventory Second Edition (BDI-II) Scoring scale at Baseline and end of study during the 8- week study period. The BDI-II Scale is a 21-item scoring tool which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represent a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe).Scores for each symptom are added up to obtain the total scores for all 21 items, which are interpreted as follows: Scores of 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression and 29-63: severe depression. The change in BDI-II scores were computed from post-intervention scores at week 8 and baseline BDI-II scores at week 0.
Time Frame: 8 weeks
Population: Only participants who completed the 8-weeks trial period were included in the final analysis of primary outcome. Per protocol analysis Post-intervention BDI-II scores at week 8 minus baseline BDI-II scores at week 0
Measure: Mean (95% Confidence Interval); unit: scores on BDI-II scale
Groups:
- Fish Oil Omega-3 EPA-rich Soft Gels Experimental Group: As the experimental group, participants received dietary supplement of OmegaVia fish oil omega-3 EPA-rich soft gels to take orally for eight weeks with bi-weekly follow-up visits. During each follow-up visit, participants were re-supplied with soft-gels and monitored for side effects and compliance.
  Each participant randomly received a sequentially numbered, securely sealed opaque plastic bottle containing fish oil omega-3 EPA-rich soft gels to take for two weeks before returning for re-supply. Three soft gels of fish oil omega-3 fatty acid were taken by each participant per day. Each soft gel contained more eicosapentaenoic acid (EPA) of 0.715 grams than docosahexaenoic acid (DHA) of 0.340 grams. The soft gels were taken orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks.
Arm/Group | Soybean Oil Soft Gels Control Group | Fish Oil Omega-3 EPA-rich Soft Gels Experimental Group
Number analyzed (Participants) | 96 | 86
scores on BDI-II scale | -13.9 [-15.3 to -12.6] | -13.3 [-14.9 to -12.0]
Statistical Analysis 1: Comparison: Soybean Oil Soft Gels Control Group vs Fish Oil Omega-3 EPA-rich Soft Gels Experimental Group; Null hypothesis: There is no difference in the magnitude of change in BDI-II scores between HIV-seropositive pregnant women on fish oil omega-3 EPA-rich supplements and the control group on soybean oil soft gels. A sample size of 91 women per arm gave an 85% power to detect as statistically significant at 5% level, a true difference of 4 scores in the mean depressive symptom scores between the two arms assuming a within group standard deviation of nine in depressive symptom scores; Test type: Superiority or Other; p = 0.21, ANCOVA — The p-value was adjusted for baseline variations in the analysis of covariance (ANCOVA) regression model. The significance level was set at p-value less than 0.05; In ANCOVA, fish oil group was main effect, participant baseline variables were covariates and presence of interaction between covariates was tested; Slope = 1.01, 95% CI 2-sided [-0.58 to 2.60], Standard Error of Mean 0.80

ADVERSE EVENTS:
Time Frame: Both known and unknown possible Adverse Events were closely monitored through out the eight-weeks study period for each participant by phone or face-to-face individual interviews and observations.
Groups:
- Soybean Oil Soft Gels: Participants on this arm received a dietary supplement of OmegaVia soybean oil soft gels as a placebo for 8 weeks with bi-weekly follow-up visits to monitor side effects and compliance.
  Soybean oil soft gels: Each participant received OmegaVia soybean oil soft gels to take orally, one soft gel taken three times per day in the morning, mid-day and in the evening after meals for a period of 8 weeks.
- Fish Oil Omega-3 EPA-rich Soft Gels: Participants received OmegaVia fish oil omega-3 EPA-rich soft gels to take orally for eight (8) weeks with bi-weekly follow-up visits for monitoring of side effects and compliance and data collection.
  Fish oil omega-3 EPA-rich soft gels: A total of 3.0g of OmegaVia fish oil omega-3 EPA-rich soft gels was taken orally per day as one soft gel in the morning, mid-day and evening after meals for 8 weeks with bi-weekly follow-up visits.
Arm/Group | Soybean Oil Soft Gels | Fish Oil Omega-3 EPA-rich Soft Gels
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/109
Other Adverse Events (participants affected / at risk) | 15/107 | 24/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Soybean Oil Soft Gels (N=107) | Fish Oil Omega-3 EPA-rich Soft Gels (N=109)
Nausea with fishy-after-taste (Gastrointestinal disorders) | 5 | 10 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Occasional vomitting in the morning after taking soft gel (Gastrointestinal disorders) | 3 | 6 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Occasional heartburn (Gastrointestinal disorders) | 5 | 3 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Occasional bloated stomach (Gastrointestinal disorders) | 0 | 2 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Occasional loose stool (Gastrointestinal disorders) | 1 | 0 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Occasional itchy skin (Skin and subcutaneous tissue disorders) | 1 | 2 — Data collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.
Nose Bleeding once (Blood and lymphatic system disorders) | 0 | 1 — This was reported only once by one participant. Data was collected throughout the 8-week study period through cell-phone regular contacts and face-to-face interviews and observations.

LIMITATIONS AND CAVEATS:
Omega-3 intake value based on international database due to absence in local food composition database. Cellular level EPA/DHA not reported due to technical problems with collected samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes